CLINICAL TRIAL: NCT05337163
Title: A Multicenter, Single-blind, Pair-matched, Observational Clinical Trial of LUNSAFE
Brief Title: A Multicenter Clinical Trial of Sputum DNA Testing for Lung Cancer in China
Status: Completed | Type: Observational
Sponsor: Creative Biosciences (Guangzhou) Co., Ltd. (Industry)
Collaborators: Guangzhou Xiangkang Medical Research Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: KLM2021-02
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer; Small Cell Lung Cancer; Non-Small Cell Lung Cancer; Squamous Cell Carcinoma; Adenocarcinoma; Large Cell Carcinoma; Adenosquamous Carcinoma; Sarcomatoid Carcinoma; Respiratory Tract Infection; Acute Bronchitis; Pneumonia; Chronic Bronchitis; Chronic Obstructive Pulmonary Disease; Tuberculosis; Lung Neoplasm; Pulmonary Interstitial Fibrosis
Keywords: Lung Cancer; Sputum DNA Test; Gene Methylation Biomarkers; Multigene Methylation Detection; Cancer Screening
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Large Cell; Carcinoma, Adenosquamous; Carcinoma; Respiratory Tract Infections; Bronchitis; Pneumonia; Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive; Tuberculosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lung cancer group: Two groups of sequential enrolled subjects, eligible subjects will be included in the study according to the inclusion criteria. In addition to collecting sputum specimen for the testing kit of Human Multigene Methylation Detection Kit (Fluorescent PCR Method) , eligible subjects also need to undergo the chest CT or pathological examination.
  Interventions: Diagnostic Test: Diagnostic Test: Sputum DNA methylation analysis; Procedure: chest CT or pathological examination
- The normal group: Two groups of sequential enrolled subjects, eligible subjects will be included in the study according to the inclusion criteria. In addition to collecting sputum specimen for the testing kit of Human Multigene Methylation Detection Kit (Fluorescent PCR Method) , eligible subjects also need to undergo the chest CT or pathological examination.
  Interventions: Diagnostic Test: Diagnostic Test: Sputum DNA methylation analysis; Procedure: chest CT or pathological examination

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Sputum DNA methylation analysis — Diagnostic Test: sputum specimen will be collected by the subject for the detection of Human Multigene Methylation Detection Kit (Fluorescent PCR Method)
  Other Names: LUNSAFE
Procedure: chest CT or pathological examination — Subjects will undergo chest CT or pathological examination.

SUMMARY:
The primary objective of this study is to assess the safety and effectiveness of Human Multigene Methylation Detection Kit (Fluorescent PCR Method) for help diagnose lung cancer by comparing with clinical standard method (includes chest CT examination or pathological examination).

DETAILED DESCRIPTION:
In this clinical trial, the testing kit to be evaluated is a Human Multigene Methylation Detection Kit (Fluorescent PCR Method), which is intended to qualitatively detect methylation levels of multiple genes in human sputum specimen in vitro by Fluorescent PCR Method, and the standard method used in clinical diagnosis is chest CT examination or pathological examination.

Subjects will provided sputum specimen as required for the evaluation of the testing kit followed by a chest CT examination or pathological examination. Technical personnel who conduct the evaluation of the testing kit will remain blinded to the results of the clinical diagnosis by chest CT and/or pathological examination.

The results of the testing kit will be compared with the standard method, and the effectiveness of the Human Multigene Methylation Detection Kit (Fluorescent PCR Method) for lung cancer detection under normal clinical use will be assessed through statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all three of the following criteria to be eligible for the study:

  1. No age or gender restrictions, voluntary participation and signing of informed consent form;
  2. Meet any of the following conditions:

  <!-- -->

  1. Suspected of lung cancer without invasive examination;
  2. Diagnosed with lung cancer without surgery, radiotherapy, chemotherapy, or targeted therapy;
  3. Diagnose other respiratory diseases, such as pulmonary infections (bacterial pneumonia, mycoplasma pneumonia, chlamydia pneumonia, viral pneumonia, lung abscess, etc.), interstitial lung diseases (pulmonary fibrosis, pulmonary granulomas, etc.), benign pulmonary nodules, tuberculosis, emphysema, pulmonary cysts, benign pulmonary tumors, obstructive pulmonary disease, bronchial infections/asthma, acute upper respiratory tract infections, etc;
  4. Diagnose other malignant tumors, such as thyroid cancer, esophageal cancer, liver cancer, gastric cancer, pancreatic cancer, etc.

Exclusion Criteria:

* Any of the following conditions must be excluded:

  1. Patients who have undergone tracheotomy or have been on a ventilator due to severe illness.
  2. The research physician believes that other reasons are not suitable for participants in this trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects without age limit, regardless of gender or region, and those who meet the inclusion criteria for this clinical trial, are eligible to enroll at the designated clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 1564 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity | One year
  Sensitivity is the percentage of subjects with lung cancer who are correctly identified by the testing kit.
Specificity | One year
  Specificity is the percentage of subjects without lung cancer who are correctly excluded by the testing kit.
Consistency Rate | One year
  Consistency rate is the fraction of both true positive and negative diagnostic test results among all subjects.
Kappa Coefficient | One year
  Kappa coefficient is the consistency analysis of the extent of agreement between the test results of the testing kit and standard method.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, PhD, Principal Investigator — Nanfang Hospital of Southern Medccal University; Laiyu Liu, PhD, Principal Investigator — Nanfang Hospital of Southern Medccal University
Locations (1):
- Nanfang Hospital of Southern Medccal University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided
  We are carefully considering all applicable regulations and laws governing sharing of patients' data from China online with the global public.